CLINICAL TRIAL: NCT06144489
Title: Plasma-Induced Changes in the Metabolome Following Polyphenol Consumption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Responsible Party: Principal Investigator, Glyn Howatson, Professor Glyn Howatson, Northumbria University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 89012
Record Dates: First submitted 2023-11-13; First posted 2023-11-22 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Processes, Metabolic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low Dose (Active Comparator): Low dose (3g) of Vistula tart cherry, freeze dried. 60-78 mg of anthocyanins, 8.07 kcal and had a macronutrient content of 1.215 g, 0.003 g, 0.042 g, for carbohydrates, fat and protein, respectively.
  Interventions: Dietary Supplement: Tart Cherry
- High Dose (Active Comparator): High dose (6g) of Vistula tart cherry, freeze dried. 120-156 mg of anthocyanins, 16.14 kcal with 2.43 g, 0.006 g, 0.08 g for carbohydrates, fat and protein, respectively.
  Interventions: Dietary Supplement: Tart Cherry
- Placebo (Placebo Comparator): Matched with the active low dose, this placebo was matched for calorific content.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Tart Cherry — Tart cherry supplementation in two doses
  Other Names: European
  Arms: High Dose; Low Dose
Dietary Supplement: Placebo — Control group
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to compare the changes in the human metabolome following a low or high acute dose of European tart cherries. The main question it aims to answer is:

what effect do European tart cherries have on the human metabolome?

Participants will attend the laboratory at the university on 3 separate occasions. Take a 3 different supplements: a placebo, low or high dose of European tart cherry supplement. Have venous blood samples taken as baseline, then 1, 2, 3, 5 and 8 h post ingestion of the supplement. Researchers will compare placebo, low and high to see if changes the human metabolome.

DETAILED DESCRIPTION:
Participants Twelve healthy participants (nine male and three female) were recruited for this study; the mean ± SD age, stature, mass and body mass index (BMI) were 29 ± 7 years old, 174.8 ± 9.3 cm, 77.29 ± 10.52 kg and 25.23 ± 1.87 kg/m2, respectively. All participants were healthy, as assessed by a health-screening questionnaire and provided written, informed consent. Exclusion criteria for the study were as follows: food allergy (as discussed with research team), history of gastrointestinal, renal, cardiovascular or thyroid disease and current use of any food supplementations. This study received ethical approval from Northumbria University Ethics Committee (reference number: 39904) (clinical trial tbc).

Experimental Design The study utilised a double blind, three-arm cross-over, pseudo-randomised (counter-balanced to eliminate order effects) design in order to identify metabolomic shifts following the acute ingestion of a low dose (LOW), high dose (HI) of TC or placebo (CON). A washout period of at least 7 days (but not greater than 21 days) between each phase was implemented. Participants were required to attend the start of each phase of the study at 7:45 am following a 10 h overnight fast in order to account for diurnal variation (Figure 1). Upon arrival to the lab, the participants baseline blood pressure (BP) was recorded in a rested state (following at least 5 mins of sitting), then cannulated for serial blood sampling. A standardized breakfast was then provided. Subsequent measures were then taken at baseline, 1, 2, 3, 5 and 8 hrs post-VTC consumption. Water was provided ad-libitum, but no additional food was given during testing visits.

Treatments and Dietary Control The low (LOW) and high (HI) dose consisted of 3 or 6 g of the TC supplement (CherryCraft), respectively, or a 3g capsule placebo (CON) matched for caloric content using maltodextrin. The low TC dose provided approximately 60-78 mg of anthocyanins, 8.07 kcal and had a macronutrient content of 1.215 g, 0.003 g, 0.042 g, for carbohydrates, fat and protein, respectively. The high TC dose provided approximately 120-156 mg of anthocyanins, 16.14 kcal with 2.43 g, 0.006 g, 0.08 g for carbohydrates, fat and protein, respectively.

Participants were requested to follow their habitual diet throughout the trial. Food diaries were completed for the 24 hrs before each testing visit to replicate (as close to) prior to testing on following testing visits. The standardized breakfast consisted of white toast (2 slices of Sainsbury's medium white bread) and butter (approx. 16g of Bertolli/Vitalite (a vegan alternative, matched as closely as possible for calories and macronutrient content)). Participants were given water to drink ad-libitum throughout the testing visits, this was measured and refilled from baseline, and 1, 2, 3, 5 and 8 hrs post breakfast and supplement ingestion.

Blood Pressure Monitoring Blood pressure was monitored throughout the testing visits, immediately upon arrival to the lab and, 1, 2, 3, 5 and 8 hrs following ingestion of the supplement.

Blood Sampling Procedure Venous blood samples (~10 mL) were collected from the antecubital fossa into lithium heparin (10 mL) tubes, immediately upon arrival to the lab and 1, 2, 3, 5 and 8 hrs following ingestion of the supplement. Samples were immediately centrifuged (3000 × g) at 4°C for 20 min, plasma was then aspirated and pipetted into ~1 mL aliquots and then immediately stored at -80 °C for later analysis.

Untargeted Plasma Analysis The sample was prepared by firstly being thawed on ice, then 200 µL of plasma was extracted and vortexed with 1000 µL of analytical grade methanol, then sonicated in a water ice bath for 15 mins. The samples were then centrifuged for 15 min at 15,000 rpm at 4°C, before the supernatant was dried in a vacuum pre-concentrator to dryness for 3 h. The residue was reconstituted in 100 µL of analytical grade water (vortex for 30 s and sonicated for 15 mins), before being filtered via 0.22 micron Costar spin filter and put in 1.5 mL autosampler vial with a 200 µL microinsert.

Metabolite characterizations were performed on a LCMS (Vanquish Liquid chromatography Front end connected to IDX High Resolution Mass Spectrometer system, Thermo Scientific, Hemel Hempstead, United Kingdom). The MS data were acquired using the AcquieX acquisition workflow (data dependent analysis). The MS operating parameters were as follows: MS1 mass resolution 60K, for MS2 30K stepped energy (HCD) 20,25,50 scan range 100-1000, RF len (%) 35, AGC gain, intensity threshold 2e4 25% custom injection mode with an injection time of 54 ms. An extraction blank was used to create a background exclusion list and a pooled QC were used to create the inclusion list. C18 RP, the chromatographic separation were archived using a Waters Acquity UPLC T3 HSS column (2.1 x 150mm with particle size of 1.7 μm), operating at 45°C with a flow rate of 200 μL/min. The LC gradient consist of binary buffer system, buffer A (LC/MS grade water/ACN 95/5 v/v) and Buffer B (LC/MS grade ACN/Water 95/5 v/v). Independent buffers system was used for positive and negative mode acquisition, the pH of buffers were adjusted using 0.1% formic acid for both. The LC gradient was the same for both polarities, 5% B at T0 hold for 1.5 min and linearly decrease to 95%B at 11min hold for 4 mins and return to starting condition and hold for further 4.5min (column stabilization). The voltage applied for positive mode was 3.5 kV and injection volume was 3 μL. The HESI condition were as follows for 200 μL: sheath gas: 35, aux gas 7 and sweep gas of 0. Ion transfer tube temperature was 300°C and vaporizer temperature was 275°C.

Data Analysis Statistical analysis was performed using SPSS (SPSS, Inc., Chicago, IL.). Descriptive statistics are reported as mean ± SD. BP was analysed using a treatment (low vs. high dose vs. placebo) by time (baseline, 1, 2, 3, 5 and 8 hrs post-supplement) repeated measures analysis of variance (RMANOVA). Mauchly's test of sphericity was used to check homogeneity of variance for all variables; where necessary, any violations of the assumption were corrected using the Greenhouse-Geisser adjustment. Significant interaction effects were followed up using post hoc analysis. The alpha level for statistical significance was set at 0.05.

ELIGIBILITY:
Inclusion Criteria:

* fit and healthy, and not currently taking any prescription medication, anti-inflammatory, anti-oxidant supplementation in the last 3 months

Exclusion Criteria:

* history of gastrointestinal, renal and/or cardiovascular disease, as well as any thyroid issues.
* smoker
* allergies
* needle/blood phobia

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2022-03-31 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-04-25 (Actual)

PRIMARY OUTCOMES:
Processes, Metabolic | up to 8 hours
  Using untargeted plasma analysis, metabolite characterisations are performed on a LCMS.

CONTACTS AND LOCATIONS:
Overall Officials: Glyn Howatson, Principal Investigator — Northumbria University
Locations (1):
- Northumbria University, Newcastle upon Tyne, Tyne and Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: No